CLINICAL TRIAL: NCT04926298
Title: Glycemic Control Before, During and After the 2016 Paris Marathon in 12 Patients With Type 1 Diabetes Using Continuous Glucose Monitoring
Brief Title: Glycemic Control Before, During and After the 2016 Paris Marathon
Acronym: MARADIAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0068
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Marathon; Physical Activity; Type 1 Diabetes Mellitus; Education; Hypoglycemia
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational mono-centric retrospective study carried out at the University Hospital of Brest The main objective of this study is to assess the glycemic control before, during and after the 2016 Paris Marathon in patients with type 1 diabetes using continuous glucose measurement (CGM) by DEXCOM sensor.

DETAILED DESCRIPTION:
Introduction

In patients with type 1 diabetes, there are general recommendations in the literature regarding carbohydrate intake and reduction of insulin doses in case of physical activity, but these recommendations should be tailored to individual patients. However, there is limited data on methods that could be applied in case of intense or extreme physical activity in patients with type 1 diabetes.

The diabetes department of Brest University Hospital has received many requests from type 1 diabetic patients for individual adaptation of insulin and carbohydrate consumption in order to participate in extreme sporting events such as marathons. One group of patients wanted to run the 2016 Paris Marathon. Our service had offered them support to define a validated method to optimize their glycemic control and prevent acute metabolic complications through 2 preparatory races preceding the Marathon de Paris 2016.

The main objective of this study is to assess the glycemic control before, during and after the 2016 Paris Marathon using continuous glucose measurement (CGM) by DEXCOM sensor.

Methods:

Study design

The study protocol consisted of 2 preparatory races (PR1 and PR2) and the Marathon. For each race, two visits were made 2 days before ("PRE" visit) and about 7 days after the race ("POST" visit).

At the first PRE visit (i.e., before PR1), patients were fitted with a DEXCOM G4® GDM device (Dexcom, San Diego, USA) to avoid a calibration problem during the periods of interest to record interstitial glycemia before, during and after each race (with calibration done in the first 24 hours). Patients were educated and trained by our care team on how to use the GCM device. Based on recommendations and our experience, patients were given advice on how to adjust their insulin therapy regimen and carbohydrate intake. In the remaining PRE visits, advice for adaptation of the insulin therapy regimen and carbohydrate intake was given to the patients based on the results of the GCM data from the previous preparatory race At the POST visit (D+7), the GCM device was removed and the GCM data was extracted using Diasend® Uploader 2.4.0 software. The GCM data was analyzed with the patient to debrief on blood glucose control during and after the race. The data was used to counsel the patient for the next race.

Preparatory race and marathon

Each patient had participated in two identical 2H preparatory races (PR1 between January and February 2016 and PR2 in March 2016). For each preparatory race, 2 or 3 groups of patients were constituted according to their physical conditions.

The Paris Marathon is a 42.195 km foot race organized every year since 1976 in the streets of Paris. On the day of the marathon, the medical and paramedical staff was divided into 3 groups. Each group was positioned at refreshment stations on the 19th, 30th and 42nd kilometers respectively.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than 3 months
* who ran the 2016 Paris Marathon;

Exclusion Criteria:

* other than type 1 diabetes;
* uncontrolled diabetes with HbA1c> 9%;
* Pregnancy;
* Coronary heart disease contraindicated for marathon running;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The therapeutic education structure of the diabetes department of the University Hospital of Brest received numerous requests from patients with type 1 diabetes for the individual tailoring of insulin and carbohydrates intake to participate in extreme sports events such as a marathon. A group of patients wished to carry out the 2016 Paris Marathon. Our department proposed to them an accompaniment to define a validated method to optimize their glycemic control and prevent acute metabolic complications through 2 preparatory races preceding the 2016 Paris Marathon
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
AUC > 200 mg/dl and <70mg/dl during Marathon | up to five days
  Area under the curve (AUC in mg/dl/min) in hyperglycemia (AUC > 200 mg/dl) and hypoglycemia (AUC < 70 mg/dl)) over 3 periods: in the 24 hours before, during and within 72 hours after the Marathon.
Time spent in hyper and hypoglycemia during Marathon | up to five hours
  Percentage of time spent with blood glucose >200mg/dl, [70-200mg/dl] and <70mg/dl) during the Marathon

SECONDARY OUTCOMES:
Insulin doses | up to five days
  Total, basal and prandial insulin doses for the periods before, during and after each run
Carbohydrate intake | up to 1 day
  Amounts of carbohydrate intake in the periods before and during each race.
AUC > 200 mg/dl and <70mg/dl during PR1 and PR2 | up to five days
  Area under the curve (AUC in mg/dl/min) in hyperglycemia (AUC > 200 mg/dl) and hypoglycemia (AUC < 70 mg/dl)) over 3 periods: in the 24 hours before, during and within 72 hours after the PR1 and PR2
Time spent in hyper and hypoglycemia during PR1 and PR2 | up to five hours
  Percentage of time spent with blood glucose >200mg/dl, [70-200mg/dl] and <70mg/dl) during the PR1 and PR2

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Brest, Brest, France